CLINICAL TRIAL: NCT05174117
Title: A Phase III Randomized Controlled Study of the Effect of Different Light Doses on Adverse Outcomes of Swallowing in Esophageal Cancer
Brief Title: Influence of Different Light Dose on the Adverse Effect of Swallowing for Esophageal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECPDT-001
Record Dates: First submitted 2021-12-21; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Esophagus Cancer
Keywords: Esophagus Cancer; Photodynamics Therapy; Laser dose
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single irradiation group (Experimental): 46-48h irradiation after photosensitizer injection: power density: 200mW·cm-2, irradiation time: 900s, volume density: 180 J·cm-2
  Interventions: Combination Product: single irradiation
- Double irradiation group (Active Comparator): 46-48h, 72h after photosensitizer injection, divided into two irradiation times: power density: 200mW·cm-2, irradiation time: 900s, volume density: 180 J·cm-2;Power density: 200mW·cm-2, irradiation time: 300s, volume density: 60 J·cm-2.
  Interventions: Combination Product: Double irradiation

INTERVENTIONS:
Combination Product: single irradiation — 46-48h irradiation after photosensitizer injection: power density: 200mW·cm-2, irradiation time: 900s, volume density: 180 J·cm-2
  Arms: single irradiation group
Combination Product: Double irradiation — 46-48h, 72h after photosensitizer injection, divided into two irradiation times: power density: 200mW·cm-2, irradiation time: 900s, volume density: 180 J·cm-2;Power density: 200mW·cm-2, irradiation time: 300s, volume density: 60 J·cm-2.
  Arms: Double irradiation group

SUMMARY:
The purpose of this experiment is to study the alleviating effects and side effects of different laser irradiation doses on esophageal stricture of esophageal cancer in order to find the appropriate dose of light.

DETAILED DESCRIPTION:
Background: Photodynamic therapy (PDT) is one of the effective means for the control of esophageal stenosis in advanced esophageal cancer, among which the dose intensity of laser irradiation is one of the factors affecting the efficacy. This study aims to pursue the appropriate dose of light.

Aim: To compare the efficacy and safety of two groups of different laser irradiation doses for advanced esophageal cancer and esophageal stricture.

Methods: Fifty-seven patients were recruited for this study and randomly divided into two groups: single irradiation group and reirradiation group.Single irradiation group: 46-48h irradiation after photosensitizer injection: power density: 200mW·cm-2, irradiation time: 900s, volume density: 180 J·cm-2;Double irradiation group: 46-48h, 72h after photosensitizer injection, divided into two irradiation times: power density: 200mW·cm-2, irradiation time: 900s, volume density: 180 J·cm-2;Power density: 200mW·cm-2, irradiation time: 300s, volume density: 60 J·cm-2.

Primary endpoints: ORR rates at 1 and 3 months, the quality of life

ELIGIBILITY:
Inclusion Criteria:

* esophagus cancer
* 18-80 years old
* grade 3-4 dysphagia （Stoller classification）
* Non-eradicative second-line treatment

Exclusion Criteria:

* Ulcerative tumor
* Esophageal stenosis caused by radiotherapy
* Survival is less than 3 months
* Patients known to be allergic to photosensitizers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
1 month objective response rate | 1 month after photodynamic irradiation
  Grade 3-4 dysphagia accounted
3 month objective response rate | 3 month after photodynamic irradiation
  Grade 3-4 dysphagia accounted

SECONDARY OUTCOMES:
3 month Quality of Life score | 3 month after photodynamic irradiation

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, MD, PhD, Study Chair — The First Affiliated Hospital of Clinical Medicine of Henan University of Science and Technology; Tanyou Shan, MD, PhD, Study Director — The First Affiliated Hospital and Clinical Medicine of Henan University of Science and Technology; Caihong Dong, MD, PhD, Principal Investigator — The First Affiliated Hospital and Clinical Medicine of Henan University of Science and Technology; Wanying Li, MD, Principal Investigator — The First Affiliated Hospital and Clinical Medicine of Henan University of Science and Technology; Jiachun Sun, MD, PhD, Principal Investigator — The First Affiliated Hospital and Clinical Medicine of Henan University of Science and Technology; Mengxi Zhang, MD, PhD, Principal Investigator — The First Affiliated Hospital and Clinical Medicine of Henan University of Science and Technology; Xiaozhi Yuan, MD, PhD, Principal Investigator — The First Affiliated Hospital and Clinical Medicine of Henan University of Science and Technology
Locations (1):
- The First Affiliated Hospital and Clinical Medicine of Henan University of Science and Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeng R, Liu C, Li L, Cai X, Chen R, Li Z. Clinical Efficacy of HiPorfin Photodynamic Therapy for Advanced Obstructive Esophageal Cancer. Technol Cancer Res Treat. 2020 Jan-Dec;19:1533033820930335. doi: 10.1177/1533033820930335. PMID 32578508
- [Background] Yoon HY, Cheon YK, Choi HJ, Shim CS. Role of photodynamic therapy in the palliation of obstructing esophageal cancer. Korean J Intern Med. 2012 Sep;27(3):278-84. doi: 10.3904/kjim.2012.27.3.278. Epub 2012 Sep 1. PMID 23019392
- [Background] Liu H, Liu Y, Wang L, Ruan X, Wang F, Xu D, Zhang J, Jia X, Liu D. Evaluation on Short-Term Therapeutic Effect of 2 Porphyrin Photosensitizer-Mediated Photodynamic Therapy for Esophageal Cancer. Technol Cancer Res Treat. 2019 Jan 1;18:1533033819831989. doi: 10.1177/1533033819831989. PMID 30885065
- [Background] Lee HH, Choi MG, Hasan T. Application of photodynamic therapy in gastrointestinal disorders: an outdated or re-emerging technique? Korean J Intern Med. 2017 Jan;32(1):1-10. doi: 10.3904/kjim.2016.200. Epub 2017 Jan 1. PMID 28049283
- [Result] Yano T, Minamide T, Takashima K, Nakajo K, Kadota T, Yoda Y. Clinical Practice of Photodynamic Therapy Using Talaporfin Sodium for Esophageal Cancer. J Clin Med. 2021 Jun 24;10(13):2785. doi: 10.3390/jcm10132785. PMID 34202917
- [Result] National Health Commission Of The People's Republic Of China. Chinese guidelines for diagnosis and treatment of esophageal carcinoma 2018 (English version). Chin J Cancer Res. 2019 Apr;31(2):223-258. doi: 10.21147/j.issn.1000-9604.2019.02.01. No abstract available. PMID 31156297